CLINICAL TRIAL: NCT04065282
Title: A Prospective, Multicenter, Single-armed, Phase II Study Evaluating Efficacy and Safety of Neoadjuvant Sintilimab in Combination With Capecitabine and Oxaliplatin (XELOX) in Patients With Resectable Locally Advanced Gastric or Gastroesophageal Adenocarcinoma.
Brief Title: The Purpose of This Study is to Evaluate the Efficacy and Safety of Sintilimab in Combination With Xelox as Neoadjuvant Therapy for Patients With Resectable Locally Advanced Gastric or Gastroesophageal Adenocarcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, jianghaiping, Associate cheif physician, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308Y030
Record Dates: First submitted 2019-08-15; First posted 2019-08-22 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Intervention Model Description: neoadjuvant chemotherapy sintilimab plus XELOX
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant therapy with Sintilimab plus Xelox (Experimental): 3 cycles of neoadjuvant therapy: Sintilimab iv d1 Q3W, Oxaliplatin 130mg/m2 iv d1 Q3W, and Capecitabine 1000mg/m2 po Bid d1-14 Q3W
  Interventions: Drug: Sintilimab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Sintilimab — 3 cycles before radical surgery
  Other Names: IBI308
Drug: Oxaliplatin — 85mg/m2 Q3W, 3 cycles perioperation
Drug: Capecitabine — 1000mg/m2 bid po D1~14 Q3W, 3 cycles perioperation

SUMMARY:
Sintilimab in Combination With Capecitabine and Oxaliplatin (XELOX) as Neoadjuvant Therapy in patients With Resectable Locally Advanced Gastric Cancer

DETAILED DESCRIPTION:
This prospective, multicenter, single-armed, phase II study will evaluate efficacy and safety of Sintilimab in combination with Xelox (Oxaliplatin 130mg/m2 iv d1 Q3w and Capecitabine 1000mg/m2 po Bid d1-14 Q3W) as neoadjuvant therapy in patients with resectable locally advanced gastric or gastroesophageal adenocarcinoma(G/GEJ AC). Newly diagnosed, treatment naïve patients with resectable locally advanced gastric or G/GEJ AC will be eligible to receive up to 3 cycles of sintilimab plus Xelox regimen as neoadjuvant therapy. Following radical gastrectomy will be performed within one to four weeks since last dosing for patients with resectable cancer after radiological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the stomach.
2. The primary tumor locates at stomach or esophagogastroesophageal ic junction.
3. Clinical T3-4NxM0 disease, confirmed by enhanced contrast abdominal computed tomography (CT) or magnetic resonance imaging (MRI).
4. At least one measurable lesion.
5. Resectable gastric or gastroesophageal cancer, judged by surgeons in this studyEligible and reasonably suitable for potentially curative resection
6. ECOG performance status 0-1.
7. Adequate organ function for chemotherapy and surgical treatment, as evaluated by laboratory tests.
8. Written (signed) informed consent.
9. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
10. Agree to use an approved contraceptive method during the treatment period, until 120 days after last dose of Sintilimab or 180 days after last dose of chemotherapy.

Exclusion Criteria:

1. Unsectable primary tumor or any distant metastatic disease.
2. Received any anti-cancer therapy for this disease, including radiation therapies, chemotherapies, immunotherapies, and Chinese traditional herb therapies.
3. Clinical T1-2N0M0 disease, confirmed by CT/MRI or endoscopic ultrasonography.
4. Active autoimmune disease or history of refractory autoimmune disease.
5. History of any other malignant tumor within 2 years, excluding cured local tumor, such as resected skin basal cell or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or ductal carcinoma in situ (DCIS).
6. History of gastrointestinal hemorrhage within 2 weeks before enrollment or patients with a high risk of hemorrhage.
7. History of gastrointestinal perforation within 6 months before enrollment.
8. Gastrointestinal obstruction, gastrointestinal dysfunction, or malabsorption syndrome that may affect the absorption of Capecitabine.
9. Weight loss is greater than 20% within 2 months before enrollment.
10. History of severe pulmonary disease, including but not limited to interstitial pulmonary disease, noninfectious pneumonitis, pulmonary fibrosis, acute pulmonary disease
11. Uncontrolled systematic disease, including diabetes mellitus, hypertension, etc.
12. Severe chronic or active infectious disease that needs systematic antibiotics, antifungal, or antiviral therapies.
13. Untreated chronic hepatitis B, serum HBV DNA load higher than the lower threshold of the test, or HCV RNA positive.
14. With any cardiovascular risk factors as follow:

    1. History of angina within 28 days before enrollment, defined as moderate pain affecting daily activities;
    2. History of symptomatic pulmonary embolism within 28 days before enrollment;
    3. History of acute myocardial infarction within 6 months before enrollment;
    4. History of NYHA class III/IV heart failure within 6 months before enrollment;
    5. History of grade 2 (Lown grading system) or menopause ventricular arrhythmias or history of supraventricular arrhythmias that needs treatment within 6 months before enrollment;
    6. History of cerebrovascular accident within 6 months before enrollment;
15. grade 1 Peripheral neuropathy , excluding patients with only deep tendon reflex absence.]
16. Known Dihydropyrimidine dehydrogenase (DPD) deficiency.
17. Known allergic to any drug used in this study.
18. History of allogeneic hematopoietic stem cell transplantation or organ transplantation.
19. Receiving corticosteroid (> 10mg/d prednisone or equivalent dose of steroids) or other systematic immunosuppression therapies within 14 days before enrollment, excluding following therapies:

    1. steroid hormone replacement therapy (≤10mg/d);
    2. local steroid therapy;
    3. short-term, prophylactic steroid therapy for preventing allergies or nausea and vomiting
20. Receiving attenuated vaccine within 4 weeks before enrollment.
21. Receiving immunotherapy or other study drugs within 28 days before enrollment,
22. History of receiving anti-PD-1, anti-PD-L1, anti-PD-L2, or any other T cell co-simulation or checkpoint inhibitor therapy.
23. Receiving major surgery within 28 days before enrollment.
24. For patients with uncontrolled epilepsy, central nervous system disease, or mental disorder, researchers should evaluate if the inform consent and/or the compliance would be affected by their disease.
25. Any drug or alcohol abuse that would affect drug management or toxicity analysis.
26. Pregnant or nursing female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | after surgical resection (up to 12 weeks after first dosing)
  evaluate pathological complete response rate of primary tumor and locally metastatic lymph nodes after 3 cycles of neoadjuvant therapy.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 9 to 12 weeks
Tumor regression grade (TRG) | after surgical resection (up to 12 weeks after first dosing)
Disease free survival (DFS) | every 90 days after resection, up to 2 years
1-year overall survival rate | 1 years
2-year overall survival rate | 2 years

OTHER OUTCOMES:
Overall survival (OS) | up to 5 years
  The relation between overall survival and pathological response after neoadjuvant therapy of Sintilimab plus Xelox for gastric cancer
PD-L1 expression, tumor infiltrating lymphocytes (TIL), etc. | after surgical resection (up to 12 weeks after first dosing)
  The relation between treatment efficacy and biomarker in tumor tissue
Cytokine (IL-6) | up to 12 weeks after first dosing
  The relation between treatment efficacy and biomarker in peripheral blood
immune cell subpopulation (CD3, CD4, CD8 lymphocytes ) | up to 12 weeks after first dosing
  The relation between treatment efficacy and biomarker in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Zhejiang, China

REFERENCES:
- [Derived] Jiang H, Yu X, Li N, Kong M, Ma Z, Zhou D, Wang W, Wang H, Wang H, He K, Li Z, Lu Y, Zhang J, Zhao K, Zhang Y, Xu N, Li Z, Liu Y, Wang Y, Wang Y, Teng L. Efficacy and safety of neoadjuvant sintilimab, oxaliplatin and capecitabine in patients with locally advanced, resectable gastric or gastroesophageal junction adenocarcinoma: early results of a phase 2 study. J Immunother Cancer. 2022 Mar;10(3):e003635. doi: 10.1136/jitc-2021-003635. PMID 35296556